CLINICAL TRIAL: NCT01047254
Title: A 12-week, Multicenter, Randomized, Double-blind, Placebo-controlled Trial of Bupropion for the Treatment of Apathy in Alzheimer's Dementia(Apa-AD)
Brief Title: Bupropion for the Treatment of Apathy in Alzheimer's Dementia
Acronym: APA-AD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Collaborators: University of Cologne (Other); Physician of neurology, psychiatry and psychotherapy Horn, MD; Bad Honnef (Unknown); Charite University, Berlin, Germany (Other); Universität Duisburg-Essen (Other); University of Erlangen-Nürnberg (Other); University of Freiburg (Other); University Medical Center Goettingen (Other); Universität des Saarlandes (Other); Johannes Gutenberg University Mainz (Other); Heidelberg University (Other); Philipps University Marburg (Other); Ludwig-Maximilians - University of Munich (Other); University of Rostock (Other); University Hospital Tuebingen (Other); University of Ulm (Other)
Responsible Party: Principal Investigator, Frank Jessen, Prof. Dr., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-005352-17
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Apathy in Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupropion (Active Comparator): Buproprion 150-300 mg in a flexible dose
  Interventions: Drug: Elontril
- placebo capsule (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Elontril — flexible dose of Bupropion 150-300 mg
  Arms: Bupropion
Drug: placebo
  Arms: placebo capsule

SUMMARY:
Apathy in dementia prevents successful application of non-pharmacological treatments, accelerates cognitive and functional decline and increases disease-related costs by earlier need for full-time care. Apathy is a distinct entity and occurs independently of other neuropsychiatric syndromes, like depression.

Today, there is no high-level evidence for any effective treatment of apathy in AD. In contrast to other neuropsychiatric syndromes in AD, like psychosis and depression, and despite its high prevalence and clinical relevance, apathy has never been the primary outcome in a clinical trial. Basic and clinical research has provided a distinct model of the pathophysiology of apathy with dopamine and norepinephrine as the key neurotransmitter systems involved. The antidepressant Bupropion is a dopamine and norepinephrine reuptake inhibitor. There is evidence from case-series, that Bupropion reduces apathy in patients with organic brain disorders. This study will test the efficacy and safety of Bupropion in the treatment of apathy in AD in a 12-week multicenter doubleblind placebo controlled trial. Secondary endpoints will be quality of life of patients, caregivers' distress, ability of patients to perform activities of daily living,utilization of healthcare resources by patients and by caregivers, and cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Alzheimer's dementia, male and female (NINCDS/ADRDA criteria)
* Presence of clinically relevant apathy defined by the Neuropsychiatric Inventory (NPI) apathy item (score of >/= 4 points) and the Marin/Starkstein criteria for apathy
* MMSE: 10-25
* Outpatient status, not institutionalized
* Presence of reliable caregiver
* Stable treatment with antidementia drugs for at least three months prior to entry or no treatment with antidementia drugs

Exclusion Criteria:

* Other Dementia (e.g. vascular dementia, Lewy-body dementia, fronto-temporal dementia)
* Presence of a clinically relevant depression defined by either the NPI depression item (score >/= 4 points) or DSM-IV criteria for major depressive episode (with depressed mood)
* Alcoholism and Benzodiazepine addiction
* Current treatment with antipsychotics and antidepressants (including St. John's wart)
* Current treatment with dopaminergic agents or Amantadin
* Current treatment with benzodiazepines
* Current treatment with MAO inhibitor (Bupropion contraindication)
* Known sensibility to Bupropion treatment
* Severe psychiatric disease (including hospitalization) in the last 6 months, suicide attempt, acute psychotic symptoms
* Severe physical illness, that do not allow a participation in a 12-week period of treatment
* Medical history with seizures
* Medical history with tumors of the central nervous system
* Severe craniocerebral injury and medical history with cerebral substance defect
* Clinically relevant renal disease, liver insufficiency
* Simultaneous treatment, which reduces the seizure threshold (e.g. antipsychotics, antidepressants, antimalarial agents, Tramadol, Theophyllin, systemic steroids in higher dose, Chinolone, sedative antihistamines)
* Simultaneous treatment, which is metabolized through Cytochrom P450-Isoenzym 2D6 (e.g. these beta blockers: Metoprolol, Proanolol, Timolol, Carvediol, Nebivolol, Typ-1C-Antiarrhyhtmics for e.g. Propafenon, Flecinid) (except Donepezil and Galantamin)
* Simultaneous treatment with drugs, which may interfere with the metabolization of Bupropion (e.g. Carbamazepin, Phenytoin, Valproat, Ritonavir, Lopinavir)
* Diabetes mellitus, which is therapeutically poorly regulated and treated by medication
* Treatment with stimulants and appetite depressants
* Participation in other clinical trials with in the last 3 months
* Suicidal tendency
* Known lactose intolerance

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in Apathy Evaluation Scale (AES) score | 12 weeks

SECONDARY OUTCOMES:
NPI total score;NPI caregivers' distress total score;ADCS-ADL; QoL-AD; RUD;ADAScog;MMSE | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jessen, MD, Principal Investigator — University Bonn
Locations (1):
- Department of Psychiatry, University Bonn, Bonn, Germany